CLINICAL TRIAL: NCT03118726
Title: Evaluation of Immediate Postpartum LARC Implementation Programs
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Lisa Hofler, Assistant Professor, University of New Mexico
Other Study IDs: 17-051
Record Dates: First submitted 2017-04-12; First posted 2017-04-18 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Post Partum Contraception
Keywords: LARC; New Mexico; Contraception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NM Perinatal Collaborative: Hospitals working with the New Mexico Perinatal Collaborative (NMPC) on implementing immediate postpartum long-acting reversible contraception programs.

SUMMARY:
This study will engage hospitals working with the New Mexico Perinatal Collaborative (NMPC) on implementing immediate postpartum long-acting reversible contraception programs. All hospitals in New Mexico interested in implementing immediate postpartum LARC programs will be eligible to participate in the NPMC program evaluation. The study will evaluate the components of this implementation program at several New Mexico hospitals using a stepped wedge design,with components being introduced to each hospital one at a time

ELIGIBILITY:
Inclusion Criteria:

* Hospital staff: Important individuals at New Mexico hospitals planning to implement immediate postpartum LARC programs, with an emphasis on diversity of administrative perspectives.
* If more than 4 potential participants are identified at one institution, additional participants may be included if their participation in the study is likely to contribute additional information (e.g. job title or background is different from other study participants)

Exclusion Criteria:

- Inability to speak and read English proficiently

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hospitals working with the New Mexico Perinatal Collaborative (NMPC) on implementing immediate postpartum long-acting reversible contraception programs. All hospitals in New Mexico interested in implementing immediate postpartum LARC programs will be eligible to participate in the NPMC program evaluation. The study will evaluate the components of this implementation program at several New Mexico hospitals using a stepped wedge design, with components being introduced to each hospital one at a time.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Baseline immediate postpartum LARC Implementation | April 2017-December 2018
  To determine baseline immediate postpartum LARC implementation in various rural New Mexico hospitals.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hofler, MD, MBA, MPH, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No